CLINICAL TRIAL: NCT02836600
Title: A Phase 1 Study of LY3039478 in Japanese Patients With Advanced Solid Tumors
Brief Title: A Study of LY3039478 in Japanese Participants With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 16191; I6F-JE-JJCC (Other: Eli Lilly and Company)
Record Dates: First submitted 2016-07-15; First posted 2016-07-19 (Estimated); Results first posted 2025-08-07 (Actual); Last update posted 2025-08-07 (Actual); Status verified 2025-07

CONDITIONS: Advanced Solid Tumor
Keywords: notch inhibitor
MeSH Terms: interventions — crenigacestat

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 25 mg LY3039478 (Experimental): Participants received 25 milligrams (mg) of LY3039478, administered orally three times per week (TIW) in a 28-day cycle, until disease progression, development of unacceptable toxicity, or any other discontinuation criteria were met.
  Interventions: Drug: LY3039478
- 50 mg LY3039478 (Experimental): Participants received 50 mg of LY3039478, administered orally TIW in a 28-day cycle, until disease progression, development of unacceptable toxicity, or any other discontinuation criteria were met.
  Interventions: Drug: LY3039478

INTERVENTIONS:
Drug: LY3039478 — Administered orally

SUMMARY:
The purpose of this study is to evaluate the tolerability of the study drug LY3039478 in Japanese participants with advanced solid tumors.

ELIGIBILITY:
Inclusion Criteria:

* Histological or cytological evidence of a diagnosis of solid tumor that is advanced and/or metastatic.
* In the judgment of the investigator, participants must be appropriate candidates for experimental therapy after available standard therapies have failed or for whom standard therapy is not appropriate.
* Performance status of less than or equal to (≤) 1 on the Eastern Cooperative Oncology Group (ECOG) scale.
* Adequate organ function, including hematologic, hepatic, and renal.
* Estimated life expectancy of greater than or equal to (≥) 12 weeks.

Exclusion Criteria:

* Received previous therapy for cancer within 14 or 21 days of the initial dose of study drug for a nonmyelosuppressive or myelosuppressive agents, respectively.
* Have serious preexisting medical conditions.
* Have current or recent (within 3 months of study drug administration) gastrointestinal disease with chronic or intermittent diarrhea.
* Have an active bacterial, fungal, and/or known viral infection.
* Have known acute or chronic leukemia or current hematologic malignancies that may affect the interpretation of results.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2016-09-09 (Actual); Primary Completion 2019-07-05 (Actual); Study Completion 2023-05-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kashiwa, Chiba, Japan

REFERENCES:
- [Derived] Doi T, Tajimi M, Mori J, Asou H, Inoue K, Benhadji KA, Naito Y. A phase 1 study of crenigacestat (LY3039478), the Notch inhibitor, in Japanese patients with advanced solid tumors. Invest New Drugs. 2021 Apr;39(2):469-476. doi: 10.1007/s10637-020-01001-5. Epub 2020 Sep 16. PMID 32939607

RESULTS

PARTICIPANT FLOW:
Recruitment Details: * This study was a dose-escalation trial that included separate groups of participants who received 25 milligrams (mg) or 50 mg of LY3039478, administered orally three times per week (TIW) in a 28-day cycle.
  * The dose was escalated from 25 mg to 50 mg only if the frequency of dose-limiting toxicity (DLT) in Cycle 1 (28 days) was less than 33 percent (<33%) among participants who had received 25 mg LY3039478.
Groups:
- 25 mg LY3039478: Participants received 25 mg of LY3039478, administered orally TIW in a 28-day cycle, until disease progression, development of unacceptable toxicity, or any other discontinuation criteria were met.
Period: Overall Study
Arm/Group | 25 mg LY3039478 | 50 mg LY3039478
Started | 4 | 7
Received at Least One Dose of LY3039478 | 4 | 7
Completed (Completers included participants who had progressive disease, died due to any cause, or were alive and on study at conclusion but off treatment.) | 4 | 7
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: All enrolled participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | 25 mg LY3039478 | 50 mg LY3039478 | Total
Number analyzed (Participants) | 4 | 7 | 11
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.25 (5.85) | 66.71 (15.10) | 65.82 (12.19)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 4
  Male | 2 | 5 | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 4 | 7 | 11
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 4 | 7 | 11
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Japan | 4 | 7 | 11

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With LY3039478 Dose-Limiting Toxicities (DLTs)
Description: DLT was defined as an adverse event (AE) that occurred during Cycle 1 (first 28 days) related to the study drug and met one of the following criteria per the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) v4.0. These criteria included: CTCAE Grade greater than or equal to (≥) 3 non-hematological toxicity, with exceptions for nausea, vomiting, or constipation, and asymptomatic electrolyte disturbances that can be controlled with standard treatment; Grade 4 hematological toxicity of greater than (>) 5 days duration; Grade ≥ 3 anemia requiring transfusion; any febrile neutropenia; neutropenia needing granulocyte-colony stimulating factors (GCSFs); Grade 3 thrombocytopenia with bleeding or requiring platelet transfusion; Grade 4 thrombocytopenia.
Time Frame: Cycle 1 (Up to 28 Days)
Population: All participants with evaluable DLT data in Cycle 1 (the first 28 days) had received greater than or equal to (≥) 75% of the assigned dose during Cycle 1 or had experienced a DLT during Cycle 1.
Measure: Count of Participants; unit: Participants
Arm/Group | 25 mg LY3039478 | 50 mg LY3039478
Number analyzed (Participants) | 4 | 6
Participants | 0 | 0

2. Secondary Outcome: Overall Response Rate (ORR): Percentage of Participants Who Achieved a Complete Response (CR) or Partial Response (PR)
Description: * The ORR was defined as the percentage of participants achieving either a CR or PR. Tumor response was assessed based on histology: Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST v1.1) was used for solid tumors, and Response Assessment in Neuro-Oncology criteria were used for glioblastoma.
  * CR was defined as the disappearance of all target lesions, with any pathological lymph nodes (whether target or non-target) showing a reduction in the short axis to <10 mm. Additionally, tumor marker results were required to have normalized. PR was defined as a decrease of at least 30% in the sum of the diameters of target lesions, using baseline diameters as the reference.
Time Frame: Baseline through Measured Progressive Disease (Up To 100 Weeks)
Population: All enrolled participants who received at least one dose of LY3039478.
Measure: Number; unit: percentage of participants
Arm/Group | 25 mg LY3039478 | 50 mg LY3039478
Number analyzed (Participants) | 4 | 7
percentage of participants
  CR | 0 | 0
  PR | 0 | 0

3. Secondary Outcome: Pharmacokinetics (PK): Maximum Observed Concentration (Cmax) of LY3039478
Description: PK: Cmax of LY3039478 was reported.
Time Frame: Cycle 1, Day 1 (Pre-dose, 0.5, 1, 2, 4, 6, 8, 10, and 24 hours post-dose); Cycle 1 Day 22 (Pre-dose, 0.5, 1, 2, 4, 6, 8, 10, and 24 hours post-dose)
Population: All enrolled participants who received at least one dose of LY3039478 and had at least one evaluable PK data. Number analyzed refer to participants evaluable at specified time points.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram per milliliter (ng/mL)
Arm/Group | 25 mg LY3039478 | 50 mg LY3039478
Number analyzed (Participants) | 4 | 7
nanogram per milliliter (ng/mL)
  Cycle 1, Day 1 | 324 (34) | 670 (39)
  Cycle 1, Day 22: number analyzed (Participants) | 3 | 4
  Cycle 1, Day 22 | 429 (69) | 416 (70)

4. Secondary Outcome: PK: Area Under the Plasma Concentration-Time Curve (AUC) From 0 to 24 Hours (AUC (0-24)) of LY3039478
Description: PK: AUC (0-24) of LY3039478 was reported.
Time Frame: as for outcome 3
Population: as for outcome 3
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms*hours per milliliter(ng*h/mL)
Arm/Group | 25 mg LY3039478 | 50 mg LY3039478
Number analyzed (Participants) | 4 | 6
nanograms*hours per milliliter(ng*h/mL)
  Cycle 1, Day 1 | 1480 (20) | 3080 (38)
  Cycle 1, Day 22: number analyzed (Participants) | 3 | 3
  Cycle 1, Day 22 | 2070 (54) | 2090 (76)

ADVERSE EVENTS:
Time Frame: Baseline to end of the follow-up (Up To 100 Weeks)
Description: All enrolled participants who received at least one dose of LY3039478.
Arm/Group | 25 mg LY3039478 | 50 mg LY3039478
All-Cause Mortality (participants affected / at risk) | 0/4 | 1/7
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/7
Other Adverse Events (participants affected / at risk) | 4/4 | 6/7
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 25 mg LY3039478 (N=4) | 50 mg LY3039478 (N=7)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Supraventricular tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Visual impairment (Eye disorders) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 3 (4)
Nausea (Gastrointestinal disorders) | 0 (0) | 3 (4)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1) | 1 (2)
Fatigue (General disorders) | 1 (1) | 0 (0)
Influenza like illness (General disorders) | 0 (0) | 1 (1)
Malaise (General disorders) | 1 (1) | 1 (1)
Pyrexia (General disorders) | 0 (0) | 1 (1)
Cystitis (Infections and infestations) | 0 (0) | 1 (1)
Lung infection (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Tinea pedis (Infections and infestations) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 0 (0) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 1 (1)
Hepatic enzyme increased (Investigations) | 2 (2) | 1 (1)
Lipase increased (Investigations) | 0 (0) | 1 (1)
Neutrophil count decreased (Investigations) | 0 (0) | 1 (2)
White blood cell count decreased (Investigations) | 0 (0) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 3 (3)
Hypophosphataemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1)
Hemiplegia (Nervous system disorders) | 1 (1) | 0 (0)
Delirium (Psychiatric disorders) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (4)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Drug eruption (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Hair colour changes (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2019-04-12): https://cdn.clinicaltrials.gov/large-docs/00/NCT02836600/Prot_000.pdf
  • Statistical Analysis Plan (2019-04-02): https://cdn.clinicaltrials.gov/large-docs/00/NCT02836600/SAP_001.pdf